CLINICAL TRIAL: NCT04013633
Title: Lowlands Saves Lives: A Randomized Trial to Assess the Impact of Face-to-face vs. Virtual Reality Training Using the Lifesaver VR-app on the Quality of Cardiopulmonary Resuscitation.
Brief Title: Lowlands Saves Lives: A Randomized Trial Comparing CPR-quality Between Face-to-face vs. Lifesaver VR Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-5422
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Out-Of-Hospital Cardiac Arrest
Keywords: Cardiopulmonary resuscitation (CPR); Basic life support (BLS); Virtual reality (VR); Education; Lay-person training
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded for study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifesaver virtual reality (VR) training (Experimental): Training using the Lifesaver VR application. Lifesaver VR is an interactive game that can be played on smartphones allowing users to 'resuscitate' a victim of cardiac arrest, while wearing VR-goggles showing a filmed CPR-scenario
  Interventions: Other: Lifesaver virtual reality training
- Face-to-face training (Active Comparator): A short face-to-face CPR training based on international guidelines provided by certified instructors
  Interventions: Other: Face-to-face training

INTERVENTIONS:
Other: Lifesaver virtual reality training — CPR training using the Lifesaver virtual reality application
  Arms: Lifesaver virtual reality (VR) training
Other: Face-to-face training — Short face-to-face CPR training
  Arms: Face-to-face training

SUMMARY:
The objective of the Lowlands Saves Lives trial is to compare the quality of cardiopulmonary resuscitation (CPR) between face-to-face versus Lifesaver Virtual Reality smartphone application trained participants using a randomized controlled trial.

DETAILED DESCRIPTION:
In order to optimize survival after out-of-hospital cardiac arrest, basic life support (BLS) training of lay-person volunteers is essential. Face-to-face training has long been considered the standard, but new training-methods have emerged, of which the Lifesaver VR (developed by the UK Resuscitation Council) app seems promising. It is unknown which training method results in the highest quality of cardiopulmonary resuscitation (CPR). Therefore, we conduct this randomized controlled trial in which subjects will be randomized to either one of the two training methods. Following the training, all participants will undergo CPR-quality testing using certified manikins and blinded assessors.

The present study will be conducted during Lowlands Science, a section of the Lowlands music festival exclusively dedicated to science. Lowlands will be held on August 16-18 of 2019 and over 50.000 attendees are expected.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years).
* Provide informed consent.

Exclusion Criteria:

* Alcohol level >0.5‰ and not able to perform tandem gait test.
* For any reason not being able to partake in the face-to-face or VR-app training (e.g. clear alcohol or drugs intoxication).
* For any reason not being able to perform the CPR test on the CPR-manikin (e.g. clear alcohol or drugs intoxication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Chest compression quality | During post-training CPR test, performed on the same day as the training
  Chest compression quality measured as depth (mm) and rate (compressions/min) measured using CPR manikin

SECONDARY OUTCOMES:
Flow fraction | During post-training CPR test, performed on the same day as the training
  Percentage of time where compressions are given, measured using CPR manikin
CPR performance score | During post-training CPR test, performed on the same day as the training
  CPR performance score from BLS-training checklist

CONTACTS AND LOCATIONS:
Overall Officials: Niels van Royen, MD, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greif R, Lockey AS, Conaghan P, Lippert A, De Vries W, Monsieurs KG; Education and implementation of resuscitation section Collaborators; Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 10. Education and implementation of resuscitation. Resuscitation. 2015 Oct;95:288-301. doi: 10.1016/j.resuscitation.2015.07.032. Epub 2015 Oct 15. No abstract available. PMID 26477418
- [Background] Bhanji F, Donoghue AJ, Wolff MS, Flores GE, Halamek LP, Berman JM, Sinz EH, Cheng A. Part 14: Education: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S561-73. doi: 10.1161/CIR.0000000000000268. No abstract available. PMID 26473002
- [Derived] Nas J, Thannhauser J, Vart P, van Geuns R, Muijsers H, Mol J, Aarts G, Konijnenberg L, Gommans D, Ahoud-Schoenmakers S, Vos JL, van Royen N, Bonnes JL, Brouwer MA. The impact of alcohol use on the quality of cardiopulmonary resuscitation among festival attendees: A prespecified analysis of a randomised trial. Resuscitation. 2022 Dec;181:12-19. doi: 10.1016/j.resuscitation.2022.10.002. Epub 2022 Oct 11. PMID 36228807
- [Derived] Nas J, Thannhauser J, Konijnenberg LSF, van Geuns RM, van Royen N, Bonnes JL, Brouwer MA. Long-term Effect of Face-to-Face vs Virtual Reality Cardiopulmonary Resuscitation (CPR) Training on Willingness to Perform CPR, Retention of Knowledge, and Dissemination of CPR Awareness: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212964. doi: 10.1001/jamanetworkopen.2022.12964. PMID 35587346
- [Derived] Nas J, Thannhauser J, van Geuns RM, van Royen N, Bonnes JL, Brouwer MA. Optimal Combination of Chest Compression Depth and Rate in Virtual Reality Resuscitation Training: A Post Hoc Analysis of the Randomized Lowlands Saves Lives Trial. J Am Heart Assoc. 2021 Jan 19;10(2):e017367. doi: 10.1161/JAHA.120.017367. Epub 2021 Jan 14. PMID 33442988
- [Derived] Nas J, Thannhauser J, Vart P, van Geuns RJ, van Royen N, Bonnes JL, Brouwer MA. Rationale and design of the Lowlands Saves Lives trial: a randomised trial to compare CPR quality and long-term attitude towards CPR performance between face-to-face and virtual reality training with the Lifesaver VR app. BMJ Open. 2019 Nov 21;9(11):e033648. doi: 10.1136/bmjopen-2019-033648. PMID 31753903
- [Derived] Nas J, Thannhauser J, Vart P, van Geuns RJ, Muijsers HEC, Mol JQ, Aarts GWA, Konijnenberg LSF, Gommans DHF, Ahoud-Schoenmakers SGAM, Vos JL, van Royen N, Bonnes JL, Brouwer MA. Effect of Face-to-Face vs Virtual Reality Training on Cardiopulmonary Resuscitation Quality: A Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):328-335. doi: 10.1001/jamacardio.2019.4992. PMID 31734702